CLINICAL TRIAL: NCT04654897
Title: A Single Dose Study to Assess the Mass Balance Recovery, Absorption, Metabolism and Excretion of [14C]-NT-814 in Healthy Male Subjects After Oral Dosing
Brief Title: Mass Balance Study of [14C]-NT-814 Oral Suspension in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21664; 2020-002987-30 (EudraCT Number)
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Open Label, single dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elinzanetant (NT-814, BAY3427080) (Experimental): Subjects received a single dose of 120 mg radioactive labeled elinzanetant ([14C]-NT-814) orally.
  Interventions: Drug: [14C]-NT-814

INTERVENTIONS:
Drug: [14C]-NT-814 — 120 mg radioactive labeled elinzanetant ([14C]-NT-814) oral suspension containing NMT (not more than) 5.6 MBq (megabecquerel) [14C].

SUMMARY:
This is a single centre, open-label, non-randomised study to assess the mass balance recovery, absorption, metabolism, and excretion of a single oral dose of [14C]-NT-814 in healthy male subjects. It is planned to enrol 6 subjects. Each subject will receive a single dose of 120 mg [14C] NT-814 containing not more than (NMT) 5.6 megabecquerel (MBq) [14C], administered as an oral suspension in the fasted state. Subjects will remain in the study until a mass balance cumulative recovery of >90% and <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 hour periods.

DETAILED DESCRIPTION:
Subjects will undergo preliminary screening procedures for the study up to 28 days before [14C]-NT-814 administration. Subjects will be admitted in the evening on the day prior to [14C]-NT-814 administration (Day -1) at which time further screening procedures will be undertaken to confirm eligibility. Subjects will be dosed in the morning of Day 1 following an overnight fast of a minimum of 8 hours.

It is planned that subjects will be released as a group when all subjects have achieved a mass balance cumulative recovery of >90% and <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 hour periods.

This may result in the subjects being discharged as a group prior to completion of the planned residency period. If the mass balance discharge criteria are achieved during the planned residency period, collection of all samples (blood, urine, and faeces) will be stopped and subjects will undergo discharge assessments. If mass balance discharge criteria have not been met by all subjects by Day 15, the residency period for the subjects not achieving the mass balance discharge criteria may be extended up to a maximum of 48 hours (i.e., up to Day 17). Blood, urine and faeces will be collected for 24 hour intervals during the extended residency period whilst the subjects are resident in the clinic.

If the mass balance discharge criteria are still not met by Day 17, subjects will enter a home collection phase during which they will collect 24-hour urine and faeces on a daily basis up until Day 24 (or until the criteria are met) and then on a weekly basis starting on Day 31 (until criteria met or Day 45 reached). During the period of weekly collection, mass balance cumulative recovery will be estimated by means of interpolation.

No additional collections will be performed for subjects who still do not meet the criteria on Day 45. Subjects entering the home collection phase will return on Day 19 ± 12 hours for blood sample collection. Discharge safety assessments will be performed at the time of actual discharge from the clinical unit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged 30 to 65 years inclusive at the time of signing informed consent.
* Body mass index (BMI) of 18.0 to 35.0 kg/m^2, inclusive, as measured at screening.
* Must be able to understand the requirement of the study and be willing to participate in the whole study.
* Must have regular bowel movements (i.e., usual stool production of ≥1 and ≤3 stools per day).
* Must provide written informed consent.
* Must agree to adhere to the contraception requirements

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1.
* Subjects who are, or are immediate family members of, a study site or Sponsor employee.
* Evidence of current SARS-CoV-2 infection.
* History of any drug or alcohol abuse in the past 2 years.
* Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type).
* A confirmed positive alcohol breath test at screening or admission.
* Current smokers and those who have smoked within the last 12 months.
* A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
* Subjects with pregnant or lactating partners.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017 [7], shall participate in the study.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the Investigator or delegate at screening.
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the Investigator.
* Subjects with biochemically verified Gilbert's Syndrome are allowed.
* Subjects with a presence of any of the following at screening, confirmed by a repeat test: AST, alanine aminotransferase or, gamma glutamyl transferase above the upper limit of normal.
* Confirmed positive drugs of abuse test result.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation.
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or GI disease, neurological or psychiatric disorder, as judged by the Investigator.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Presence or history of clinically significant allergy requiring treatment, as judged by the Investigator.
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood.
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) in the 14 days before IMP administration.
* History of GI surgery (with the exception of appendectomy unless it was performed within the previous 3 months).
* Acute diarrhoea or constipation in the 7 days before the predicted Day 1.
* Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Mass Balance Recovery of Total Radioactivity: CumAe(Urine) | Day 45 (maximum)
  CumAe(Urine): cumulative amount of Total Radioactivity (TR) excreted in urine.
Mass Balance Recovery of Total Radioactivity: Cum%Ae(Urine) | Day 45 (maximum)
  Cum%Ae(Urine): cumulative amount of TR excreted in urine expressed as a percentage of the radioactive dose administered.
Mass Balance Recovery of Total Radioactivity: CumAe(Faeces) | Day 45 (maximum)
  CumAe(Faeces): cumulative amount of TR excreted in faeces.
Mass Balance Recovery of Total Radioactivity: Cum%Ae(Faeces) | Day 45 (maximum)
  Cum%Ae(Faeces): cumulative amount of TR excreted in faeces expressed as a percentage of the radioactive dose administered.
Mass Balance Recovery of Total Radioactivity: CumAe(Total) | Day 45 (maximum)
  CumAe(Total): cumulative amount of TR excreted in urine and faeces combined. The radioactivity associated with toilet tissue was also determined, and the results were reported for each subject as a single value for the whole collection period only and included in the calculation of total Ae and % of dose recovered. The data reported for total calculations excluded toilet tissue data for the 0 - 6 hours post-dose to 0 - 456 hours post-dose collection intervals and included toilet tissue data for the 0 - 480 hours post-dose collection interval.
Mass Balance Recovery of Total Radioactivity: Cum%Ae(Total) | Day 45 (maximum)
  Cum%Ae(Total): cumulative amount of TR excreted in urine and faeces combined expressed as a percentage of the radioactive dose administered. The radioactivity associated with toilet tissue was also determined, and the results were reported for each subject as a single value for the whole collection period only and included in the calculation of total Ae and % of dose recovered. The data reported for total calculations excluded toilet tissue data for the 0 - 6 hours post-dose to 0 - 456 hours post-dose collection intervals and included toilet tissue data for the 0 - 480 hours post-dose collection interval.

SECONDARY OUTCOMES:
AUC(0-tlast) of NT-814 (in plasma) | Day 45 (maximum)
  AUC(0-tlast): Area under the curve from time 0 to the time of last measurable concentration.
AUC(0-tlast) of Total Radioactivity (in plasma and whole blood) | Day 45 (maximum)
  AUC(0-tlast): Area under the curve from time 0 to the time of last measurable concentration.
Cmax of NT-814 (in plasma) | Day 45 (maximum)
  Cmax: Maximum observed concentration.
Cmax of Total Radioactivity (in plasma and whole blood) | Day 45 (maximum)
  Cmax: Maximum observed concentration.
Ae(urine) by interval | Day 45 (maximum)
  Ae(urine): amount of TR excreted in urine.
%Ae(urine) by interval | Day 45 (maximum)
  %Ae(urine): amount of TR excreted in urine expressed as a percentage of the radioactive dose administered.
Ae(faeces) by interval | Day 45 (maximum)
  Ae(faeces): amount of TR excreted in faeces.
%Ae(faeces) by interval | Day 45 (maximum)
  %Ae(faeces): amount of TR excreted in faeces expressed as a percentage of the radioactive dose administered.
Ae(total) by interval | Day 45 (maximum)
  Ae(total): amount of TR excreted in urine and faeces combined.
%Ae(total) by interval | Day 45 (maximum)
  %Ae(total): amount of TR excreted in urine and faeces combined expressed as a percentage of the radioactive dose administered.
CumAe(urine) by interval | Day 45 (maximum)
  CumAe(urine): cumulative amount of TR excreted in urine.
%CumAe(urine) by interval | Day 45 (maximum)
  %CumAe(urine): cumulative amount of TR excreted in urine expressed as a percentage of the radioactive dose administered.
CumAe(faeces) by interval | Day 45 (maximum)
  CumAe(faeces): cumulative amount of TR excreted in faeces.
%CumAe(faeces) by interval | Day 45 (maximum)
  %CumAe(faeces): cumulative amount of TR excreted in faeces expressed as a percentage of the radioactive dose administered.
CumAe(total) by interval | Day 45 (maximum)
  CumAe(total): cumulative amount of TR excreted in urine and faeces combined. H=hour. The radioactivity associated with toilet tissue was also determined, and the results were reported for each subject as a single value for the whole collection period only and included in the calculation of total Ae and % of dose recovered. The data reported for total calculations excluded toilet tissue data for the 0 - 6 hours post-dose to 0 - 456 hours post-dose collection intervals and included toilet tissue data for the 0 - 480 hours post-dose collection interval.
%CumAe(total) by interval | Day 45 (maximum)
  %CumAe(total): cumulative amount of TR excreted in urine and faeces combined expressed as a percentage of the radioactive dose administered. H=hour. The radioactivity associated with toilet tissue was also determined, and the results were reported for each subject as a single value for the whole collection period only and included in the calculation of total Ae and % of dose recovered. The data reported for total calculations excluded toilet tissue data for the 0 - 6 hours post-dose to 0 - 456 hours post-dose collection intervals and included toilet tissue data for the 0 - 480 hours post-dose collection interval.
Evaluation of the extent of distribution of Total Radioactivity (TR) into blood cells | Up to 45 days
  Plasma concentration ratios for TR is reported.
Number of subjects with treatment-emergent adverse events | Up to 45 days
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation subject that does not necessarily have a causal relationship with treatment. Treatment-emergent AEs are AEs that commenced during/after the administration of investigational medicinal product (IMP) or commenced before administration of IMP (i.e., a pre-dose AE or existing medical condition) but worsened in intensity during exposure to IMP.
Laboratory Evaluations - number of subjects with clinically important changes in hematology and clinical chemistry parameters from baseline | Baseline, 24 hours post-baseline and at Discharge
Vital Signs - number of subjects with clinically important changes in systolic and diastolic blood pressure and heart rate from baseline | Baseline, 1 hour, 4 hours, 24 hours post-baseline and at Discharge
Number of subjects with clinically relevant findings in electrocardiogram (ECG) parameters from baseline | Baseline, 1 hour, 4 hours, 24 hours post-baseline and at Discharge
Number of subjects with clinically significant abnormal findings in physical examination | Up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Prinicipal Investigator, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Schulz SI, Schultze-Mosgau MH, Engelen A, Singh N, Pawsey S, Francke K, Lock R, Rottmann A. Mass Balance Recovery, Absorption, Metabolism, and Excretion of Elinzanetant in Healthy Human Volunteers and in vitro Biotransformation. Eur J Drug Metab Pharmacokinet. 2025 Jan;50(1):91-103. doi: 10.1007/s13318-024-00930-3. Epub 2024 Dec 24. PMID 39719488
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/